CLINICAL TRIAL: NCT03076489
Title: Hed-O-Shift: Hedonic and Neurocognitive Processes in Relation to Dietary Habits and Weight Status
Acronym: Hed-O-Shift
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 35RC17_9740_Hed-O-Shift
Record Dates: First submitted 2017-03-07; First posted 2017-03-10 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Neurocognitive Correlates of Eating Habits
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high consumption habits (Experimental): high consumption habits of fatty and sugary foods
  Interventions: Other: First Visit; Other: on-line questionnaires; Device: fMRI
- low consumption habits (Experimental): low consumption habits of fatty and sugary foods
  Interventions: Other: First Visit; Other: on-line questionnaires; Device: fMRI

INTERVENTIONS:
Other: First Visit — blood sample , morpho-anatomic measures (height, weight, hip and size), impedancemetry and resting energy expenditure by indirect calorimetry, sample of urine and faeces previously collected at home
Other: on-line questionnaires — The two on-line questionnaires (hedonic and caloric evaluation of foods and beverages on photos) will have to be completed by the volunteers between the first and the second visit to the University-Hospital.
Device: fMRI — a cognitive two-choice test based on food and drink pictures, during fMRI. Before and after the fMRI session, an assessment of the state of hunger, thirst, and general status of the volunteer will be carried out using a numerical scale ranging from 1 to 10.

SUMMARY:
This study includes an inclusion visit, 2 visits to the Rennes University Hospital and the filling of two on-line questionnaires.

The first visit to the University-Hospital of Rennes, during which a blood sample will be taken, morpho-anatomic measures (height, weight, hip and size), impedancemetry and resting energy expenditure by indirect calorimetry will be carried out in the Clinical Investigation Unit.

During this visit, the volunteers will also have to bring a sample of urine and faeces previously collected at home.

The two on-line questionnaires (hedonic and caloric evaluation of foods and beverages on photos) will have to be completed by the volunteers between the first and the second visit to the University-Hospital.

Finally, the volunteers will go to the University-Hospital of Rennes for the second visit, on the Neurinfo platform, during which they will be subjected to a cognitive two-choice test based on food and drink pictures, during fMRI. Before and after the fMRI session, an assessment of the state of hunger, thirst, and general status of the volunteer will be carried out using a numerical scale ranging from 1 to 10.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-24,
* Presenting a normal BMI (18-25),
* Right-handers,
* Affiliated to a social security scheme
* Having given a free, informed and written consent.
* Having a low frequency of consumption of fatty and / or sugary / salty foods, or on the contrary, a high frequency of consumption of these foods.

Exclusion Criteria:

* Related to the study:
* High level athletes, (determined on the basis of the Ricci & Gagnon questionnaire - excluded if score > 32);
* Food abstinents for religious, ideological or health reasons (intolerance, vegetarianism, allergies, etc.);
* Family history of obesity or diabetes;
* Personal history of TCA, anxiety or depressive disorder, or proven addictive behaviour;
* Excessive consumption of alcohol or other psychoactive substances (determined on the basis of the AUDIT questionnaires - excluded if score > 7 and CRAFT - excluded if score> 2 " yes ");
* Smoking daily or having stopped for less than 6 months;
* History of bariatric surgery;
* On-going treatment in the nutrition unit;
* Insufficient command of French;
* Pregnant or nursing women;
* Persons of full age who are subject to legal protection (safeguard of justice, curatorship, guardianship), persons deprived of their liberty.
* Simultaneous participation in another research protocol involving the human person

Related to fMRI:

* Implantable cardiac pacemaker or defibrillator;
* Neurosurgical clips;
* Cochlear implants;
* Neural or peripheral stimulator;
* Foreign orbital or brain metallic foreign bodies;
* Endoprostheses implanted for less than 4 weeks and osteosynthesis materials placed for less than 6 weeks;
* Claustrophobia.

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
Significant change in cerebral activity in zones involved in food intake inhibition control | at 2 weeks
  Significant change in cerebral activity (expressed as a significant variation in hemodynamic response BOLD in the condition of food cognitive tasks) in zones involved in food intake inhibition control (dorso-lateral prefrontal cortex, upper frontal gyrus)

SECONDARY OUTCOMES:
Significant change in cerebral activity in areas involved in the control of reward and motivation (striatum dorsal, insula), associated with modulation of the intestinal microbiota and metabolic and hormonal homeostasis. | at 2 weeks
  Significant change in cerebral activity in areas involved in the control of reward and motivation (striatum dorsal, insula), associated with modulation of the intestinal microbiota and metabolic and hormonal homeostasis.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Rennes Pontchaillou, Rennes, France

REFERENCES:
- [Result] Constant A, Gautier Y, Coquery N, Thibault R, Moirand R, Val-Laillet D. Emotional overeating is common and negatively associated with alcohol use in normal-weight female university students. Appetite. 2018 Oct 1;129:186-191. doi: 10.1016/j.appet.2018.07.012. Epub 2018 Jul 17. PMID 30009932
- [Result] Coquery N, Gautier Y, Serrand Y, Meurice P, Bannier E, Thibault R, Constant A, Moirand R, Val-Laillet D. Brain Responses to Food Choices and Decisions Depend on Individual Hedonic Profiles and Eating Habits in Healthy Young Women. Front Nutr. 2022 Jun 24;9:920170. doi: 10.3389/fnut.2022.920170. eCollection 2022. PMID 35811938